CLINICAL TRIAL: NCT02443779
Title: Relationship Between Symptom Severity, Retinal Morphology, and the Nigrostriatal Dopamine System in the Brain in Parkinson's Disease
Brief Title: Relationship Between Symptoms, Retinal Morphology, and the Nigrostriatal Dopamine System in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Wills Eye Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15D.060
Record Dates: First submitted 2015-04-30; First posted 2015-05-14 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Parkinson's disease patients: All subjects will undergo a complete neuro-ophthalmological examination, including assessment of best-corrected visual acuity, ocular motility, pupillary reflexes, slit-lamp biomicroscopy, intraocular pressure (IOP) measurement, and dilated fundus examination, followed by an optical coherence tomography study. Subjects will also have a DaTscan for striatal dopamine transporter visualization using single photon emission computed tomography (SPECT) brain imaging. A clinical examination will also be performed in order to document motor and cognitive functioning.
- Advanced Parkinson's disease patients: All subjects will undergo a complete neuro-ophthalmological examination, including assessment of best-corrected visual acuity, ocular motility, pupillary reflexes, slit-lamp biomicroscopy, intraocular pressure (IOP) measurement, and dilated fundus examination, followed by an optical coherence tomography study. Subjects will also have a DaTscan for striatal dopamine transporter visualization using single photon emission computed tomography (SPECT) brain imaging. A clinical examination will also be performed in order to document motor and cognitive functioning.

SUMMARY:
The purpose of this study is to examine if a correlation exists between findings from brain imaging studies of the status of the dopamine system in the brain using DaTscan and SPECT imaging, clinical symptoms of Parkinson's disease, and changes in the structure of the retina as detected by optical coherence tomography (OCT) in recently diagnosed and more advanced Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Between the ages of 50-80 years old.
3. Male or female with idiopathic PD who fulfill UK PD Society brain bank criteria for diagnosis of Parkinson's disease.
4. Early stage subjects will need to have Unified Parkinson's Disease Rating Scale (UPDRS) motor scores of < 10, be within 3 years of diagnosis, and not requiring dopaminergic therapy
5. Later stage subjects will need to have Unified Parkinson's Disease Rating Scale motor scores of > 20 and be > 5 years from diagnosis
6. If female, one of the following three scenarios must apply:

   * at least two years post-menopausal
   * surgically sterile
   * negative urine pregnancy test, and following a reliable method of birth control (oral contraceptive, intrauterine device, contraceptive implant, barrier, or abstinence) for at least two months prior to entry, and agreeing both to follow a reliable method of birth control, and (if relevant) to desist from breast feeding during, and for two weeks following tracer administration.

Exclusion Criteria:

1. Abrupt onset of Parkinsonism
2. 'Other Parkinson-like syndromes (e.g. progressive supranuclear palsy, multiple system atrophy)
3. Any condition that would preclude successful completion of SPECT scanning
4. Use of anti-coagulant therapy
5. Any clinically significant eye disease that would complicate interpretation of OCT data
6. Use of any drugs that would alter or interfere with tracer binding for SPECT imaging studies (ex., cocaine, amphetamines, methylphenidate, ephedrine, phentermine, bupropion, fentanyl, selective serotonin reuptake inhibitors).
7. Known sensitivity to the imaging agent or to Lugol's solution or to potassium perchlorate.
8. History or presence of severe renal disease.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be Parkinson's disease patients (Hoehn and Yahr stage 1 - 3). One study group will be subjects (N = 6) with early PD who will be within 3 years from diagnosis and not requiring dopaminergic therapy. These subjects will need to have Unified Parkinson's Disease Rating Scale motor scores of 10 - 15. The second study group will be subjects (N = 6) with more advanced PD and will have had PD for at least 5 years and will need to have Unified Parkinson's Disease Rating Scale motor scores of > 20.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-12; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
OCT results | 1 day
  OCT measures including measurements of the thickness (microns) of specific retinal layers including RNFL, ganglion cell layer, inner plexiform layer, inner nuclear layer, outer plexiform layer, outer nuclear layer, photoreceptors, and retinal pigment epithelium.
DaTscan results | 1 day
  Striatal binding ratios will be calculated for striatal regions of interest.
Clinical examination results | 1 day
  UPDRS motor score

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Schneider, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States